CLINICAL TRIAL: NCT04360382
Title: Enhanced Recovery Versus Conventional Care After Cesarean Section: Role Of Nursing
Brief Title: Enhanced Recovery Versus Conventional Care After Cesarean Section
Status: Completed | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: IRB approval number.258691
Record Dates: First submitted 2020-02-15; First posted 2020-04-24 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cesarean Section; Enhanced Recovery
Keywords: cesarean section; Nursing; Enhanced recovery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enhanced recovery: Part I: Preoperative evaluation and preparation:
  Part II: Postoperative daily intervention:
  Part III: Expected daily outcome :
  Phase three: Implementing enhanced recovery program:
  The established pathway will implement on the study group by researcher from admission till discharge as conventional care group assessment in phase one.
  Phase four: Evaluating enhanced recovery program outcomes:
  The efficacy of enhanced recovery program will be determined by comparing outcomes for patients of both control and study groups
  Interventions: Other: ERACS; Other: Regular care
- Regular care: usual care for all cases of cesarean section at our hospital.
  Interventions: Other: ERACS; Other: Regular care

INTERVENTIONS:
Other: ERACS — Pregnant women scheduled for cesarean section will be subjected to preoperative, intra-operative and postoperative nurse care aiming at early recovery.
Other: Regular care — Usual care for all cases subjected to cesarean section at our hospital.

SUMMARY:
A protocol of ERACS is introduced to our hospital aiming at saving a lot of time and money for the patients and the population at large .By this way ,free beds for more cases can be available for others patients, so the researcher is welling to study this research on women undergoing CS at Woman's Health University Hospital.

DETAILED DESCRIPTION:
This study aims to assess the level of satisfaction of the women undergoing Enhanced Recovery Program (ERP) versus conventional care after cesarean section..

The study will be conducted at the woman's Health University Hospital at obstetrics ward and postpartum ward of that hospital,at the Assuit

The sample size for this study will be 300 randomized -controlled trails women and divided into two groups :

The first 150 of women will be enrolled to the control group, receiving conventional care and the second 150 of women will be recruited to the study group , receiving enhanced recovery program based care .

* Randomization will done by using computer -generated random table.
* After acceptance of eligible women to participate in the study ,they will assigned randomly to either one of the above groups.

Two tools will be used to collect data of this study:

Tool I: perioperative cesarean Section assessment tool:

This tool will be developed by the researcher based on reviewing available related literature and will be used to collect data regarding outcomes .

This tool will include the following parts:

Part 1:women's personal data: Consisted of 6 questions such as age, level of education , occupation, weight, height, indication for CS ,date ,time of admission and discharge .

Part 2: preoperative Data: Consisted of 13 questions such as present medical ,past and surgical histories, obstetric history ,smoking history , vital signs, investigations, patient advice and information ,breast feeding education ,discuss NPO status (reduced fasting times ),hemoglobin optimization ,contact women the day before delivery to review ERAS goals , bowel preparation, ,medications, time of transfer to theatre.

Part 3:Intraopreative Data: Consisted of 10 questions such as duration of operation , total fluid replacement ( including blood transfusion), vital signs ,urine output ,active warming, delayed cord clamping , skin to skin contact on operation table , minimally invasive surgical technique, anesthetic and analgesia medication .

Part 4:Post-operative Data: Consisted of 16 questions such as time of admission to ward, time of starting oral fluid, time of mobilization , time of remove urinary catheter ,duration of IV fluid ,use of chewing gum in early postoperative period ,pain intensity , use of analgesia drug and anibiotics,postoperative complication, pain intensity on discharge ,postoperative length of stay and reason of delayed postoperative length of stay.

Tool II: Patient's satisfaction tool:

This tool will be developed by researcher based on reviewing related literature including existing satisfaction tools, tested of validity ,piloted for internal consistency reliability ,scored and will utilize to assess patient's satisfaction about quality of perioperative care services. It is six domains and 40 items. Hospital admission procedure domain ( has 4 domains) such as women satisfied about ease of overall ,health care domain (has 10 domains) such as women satisfied about number of around made of doctor, physician services ,information provision domain (has 13 domains) such as women satisfied about information of breast feeding and pain management , ,the personal treatment domain (has 5 domains) such as women satisfied about kindness of staff , food domain (has 3 domains) such as women satisfied about served food quality (has 5 domains) such as women satisfied about cleanliness in the room and hospital facilities .

- Patient's satisfaction will measures by using four points Likert's scale ; Four point Likert's format that goes from strongly satisfied (4) to strongly dissatisfied (1), which helps in obtaining an ordinal measure of the strength of the satisfaction with each item. The tool score range from 40 to 160 .The score of ≤ 80 = dissatisfied, the range score > 80- 120 = satisfied , and the range score of > 120 - 160 = very satisfied (Ahmed et.al,2017).

Validity of data collection tools Content validity of the data collection tools will be established by 5 experts in the field of the study .The necessary modifications will be done accordingly.

Pilot study:

A pilot study will be carried out on the first 10 % of the total sample to test the content validity, feasibility, clarity and objectively of the tool as well as estimate the time needed for data collection. Data will analyzed manually following pilot study. According to the result of pilot study the necessary modifications will be done accordingly.

procedure: An written official approval letter from Faculty of Nursing at the University of Assuit to the director of Women Health Hospital; this letter will include a brief explanation of the objective and permission to carry out the study .

Data will be collected from control group first and then from study group to prevent sample contamination. The control group will receive the conventional care while study group will receive developed enhanced recovery program care .

Phase 1: Conventional Care Assessment Perioperative data will be collected from this group by tool I .Every patient will be assessed at a day before operation to gather all preoperative data .the women's operative report is reviewed by researcher and required information will be recorded on data collection tool .After that women will be followed up till she is transferred to postpartum ward where patient will daily be reassessed during morning shift till patient discharge. The patient's satisfaction will be assessed at discharge using tool II .

Phase 2: Designing enhanced recovery program:

Based on reviewing related to literature; enhanced recovery program after cesarean section will be formulated by a designer team, which will consist of a supervisor and head nurse of ward, and researcher.

The established enhanced recovery pogram will consist of four parts:

Part I: Preoperative evaluation and preparation:

This part will include health history, physical examination, and diagnostic investigation, as well as pre-operative patient preparation.

Part II: Postoperative daily intervention:

This part will include the daily nursing and collaborative interventions such as assessment, nutrition, activities, medications, patient and family education, and discharge planning and instructions.

Part III: Expected daily outcome :

This part will include the patient's daily outcomes such as vital signs stability , pain control ,activities of daily living and mobility improvement; return bowel function, and meeting discharge criteria .

Phase three: Implementing enhanced recovery program:

The established pathway will implement on the study group by researcher from admission till discharge as conventional care group assessment in phase one.

Phase four: Evaluating enhanced recovery program outcomes:

The efficacy of enhanced recovery program will be determined by comparing outcomes for patients of both control and study groups

ELIGIBILITY:
Inclusion Criteria:

* Women from 20- 40 years old .
* Women Undergoing elective cesarean Section.
* Low risk pregnancy; no medical ,surgical or obstetric problem.

Exclusion Criteria:

* Emergency cesarean section.
* Women who refuse to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Elective cesarean section for a pregnany woman.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative length of hospital stays of stay. | 1 week
  Hospital stay after CS in hours. The shorter stay is the better.
Breast feeding initiation | 1 month
  Physiologic scale: Amount and onset of milk secretion. The sufficient amount with early lactation is the better.
Pain control | 1 month
  Visual analogue pain scale. Minimal or low pain is the better.

SECONDARY OUTCOMES:
Financial cost score | 1 month
  The less cost is the better.

CONTACTS AND LOCATIONS:
Overall Officials: Atef Darwish, Principal Investigator — Woman's Health University Hospital
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided